CLINICAL TRIAL: NCT02768597
Title: A Prospective, Randomized Study Comparing The Outcome of Large-Diameter vs Small-Diameter Glenospheres in Primary Reverse Shoulder Arthroplasty Using the ReUnion System
Brief Title: Comparing The Outcome of Large-Diameter vs Small-Diameter Glenospheres in Primary Reverse Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Principal Investigator, Mark E. Morrey, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-006839
Record Dates: First submitted 2016-04-20; First posted 2016-05-11 (Estimated); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Glenohumeral Joint Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Large-Diameter Glenosphere +2 mm offset (Active Comparator): Primary Reverse Shoulder Arthroplasty using the ReUnion System with a Large-Diameter Glenosphere +2 mm offset
  Interventions: Device: ReUnion System with a Large-Diameter Glenosphere +2 mm offset
- Small-Diameter Glenosphere +2 mm offset (Active Comparator): Primary Reverse Shoulder Arthroplasty using the ReUnion System with a Small-Diameter Glenosphere +2 mm offset
  Interventions: Device: ReUnion System with a Small-Diameter Glenosphere +2 mm offset
- Large-Diameter Glenosphere +6 mm offset (Active Comparator): Primary Reverse Shoulder Arthroplasty using the ReUnion System with a Large-Diameter Glenosphere +6 mm offset
  Interventions: Device: ReUnion System with a Large-Diameter Glenosphere +6 mm offset
- Small-Diameter Glenosphere +6 mm offset (Active Comparator): Primary Reverse Shoulder Arthroplasty using the ReUnion System with a Small-Diameter Glenosphere +6 mm offset
  Interventions: Device: ReUnion System with a Small-Diameter Glenosphere +6 mm offset

INTERVENTIONS:
Device: ReUnion System with a Large-Diameter Glenosphere +2 mm offset — Primary Reverse Shoulder Arthroplasty using the ReUnion System with a Large-Diameter Glenosphere +2 mm offset
  Arms: Large-Diameter Glenosphere +2 mm offset
Device: ReUnion System with a Small-Diameter Glenosphere +2 mm offset — Primary Reverse Shoulder Arthroplasty using the ReUnion System with a Small-Diameter Glenosphere +2 mm offset
  Arms: Small-Diameter Glenosphere +2 mm offset
Device: ReUnion System with a Large-Diameter Glenosphere +6 mm offset — Primary Reverse Shoulder Arthroplasty using the ReUnion System with a Large-Diameter Glenosphere +6 mm offset
  Arms: Large-Diameter Glenosphere +6 mm offset
Device: ReUnion System with a Small-Diameter Glenosphere +6 mm offset — Primary Reverse Shoulder Arthroplasty using the ReUnion System with a Small-Diameter Glenosphere +6 mm offset
  Arms: Small-Diameter Glenosphere +6 mm offset

SUMMARY:
The study will compare the outcome of primary reverse shoulder arthroplasty using the Stryker ReUnion System with implantation of either a large (40 mm) or a small (36 mm) glenosphere with either a +2 mm or a +6 mm offset.

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to sign the informed consent
* Male and non-pregnant female subjects ages 50 - 90 at the time of surgery
* Subjects requiring a primary reverse total shoulder arthroplasty
* Subjects with the diagnosis of cuff-tear arthropathy (CTA), massive irreparable rotator cuff tear (MRCT) or osteoarthritis (OA) with marked posterior subluxation or bone loss

Exclusion Criteria:

* Inability to comply with follow-up requirements
* Subjects with inflammatory arthritis
* Subjects with proximal humerus fractures
* Subjects with sequels of trauma
* Subjects that are immunologically compromised
* Subjects with an active or suspected latent infection in or about the shoulder
* Need to add a tendon transfer
* Need for structural humeral bone graft
* Pregnant subjects

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2016-04; Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Morrey, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
Started | 34 | 28 | 29 | 22
Completed | 34 | 28 | 29 | 22
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset | Total
Number analyzed (Participants) | 34 | 28 | 29 | 22 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.65 (8.24) | 72.90 (7.92) | 73.75 (7.20) | 71.98 (7.72) | 72.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 15 | 8 | 55
  Male | 16 | 14 | 14 | 14 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 34 | 28 | 29 | 22 | 113

OUTCOME MEASURES:

1. Primary Outcome: Active Forward Elevation of the Shoulder
Description: Degrees of movement the participant is able to independently lift arm upward to the ceiling, while keeping elbow straight. Normal movement for forward elevation is 180 degrees.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: degrees of movement
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
Number analyzed (Participants) | 34 | 28 | 29 | 22
degrees of movement | 146 (15) | 141 (28) | 143 (19) | 137 (20)
Statistical Analysis 1: Comparison: Small-Diameter Glenosphere +2 mm Offset vs Small-Diameter Glenosphere +6 mm Offset vs Large-Diameter Glenosphere +2 mm Offset vs Large-Diameter Glenosphere +6 mm Offset; Test type: Superiority; p = .552, ANOVA

2. Primary Outcome: Active External Rotation of the Shoulder
Description: Degrees of movement the participant is able to independently rotate arm up, while keeping arm at 0 degrees of abduction. Normal movement for external rotation is 90 degrees.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: degrees of movement
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
Number analyzed (Participants) | 34 | 28 | 29 | 22
degrees of movement | 55 (17) | 60 (18) | 52 (22) | 54 (17)
Statistical Analysis 1: Comparison: Small-Diameter Glenosphere +2 mm Offset vs Small-Diameter Glenosphere +6 mm Offset vs Large-Diameter Glenosphere +2 mm Offset vs Large-Diameter Glenosphere +6 mm Offset; Test type: Superiority; p = .558, ANOVA

3. Primary Outcome: Shoulder Abduction Strength
Description: Shoulder abduction strength was measured using manual testing where strength was graded as: (1) paralysis; (2) contraction with no ability to resist gravity; (3) weak but able to resist gravity; (4) weak but able to resist the examiner; (5) normal.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
Number analyzed (Participants) | 34 | 28 | 29 | 22
units on a scale | 4.8 (0.4) | 4.5 (0.6) | 4.7 (0.5) | 4.8 (0.4)
Statistical Analysis 1: Comparison: Small-Diameter Glenosphere +2 mm Offset vs Small-Diameter Glenosphere +6 mm Offset vs Large-Diameter Glenosphere +2 mm Offset vs Large-Diameter Glenosphere +6 mm Offset; Test type: Superiority; p = .274, Kruskal-Wallis

4. Primary Outcome: Shoulder External Rotation Strength
Description: Shoulder external rotation strength was measured using manual testing where strength was graded as: (1) paralysis; (2) contraction with no ability to resist gravity; (3) weak but able to resist gravity; (4) weak but able to resist the examiner; (5) normal.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
Number analyzed (Participants) | 34 | 28 | 29 | 22
units on a scale | 4.8 (0.4) | 4.6 (0.6) | 4.7 (0.5) | 4.7 (0.4)
Statistical Analysis 1: Comparison: Small-Diameter Glenosphere +2 mm Offset vs Small-Diameter Glenosphere +6 mm Offset vs Large-Diameter Glenosphere +2 mm Offset vs Large-Diameter Glenosphere +6 mm Offset; Test type: Superiority; p = .539, Kruskal-Wallis

5. Primary Outcome: Shoulder Internal Rotation Strength
Description: Shoulder internal rotation strength was measured using manual testing where strength was graded as: (1) paralysis; (2) contraction with no ability to resist gravity; (3) weak but able to resist gravity; (4) weak but able to resist the examiner; (5) normal.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
Number analyzed (Participants) | 34 | 28 | 29 | 22
units on a scale | 4.9 (0.3) | 4.8 (0.4) | 4.7 (0.4) | 4.9 (0.3)
Statistical Analysis 1: Comparison: Small-Diameter Glenosphere +2 mm Offset vs Small-Diameter Glenosphere +6 mm Offset vs Large-Diameter Glenosphere +2 mm Offset vs Large-Diameter Glenosphere +6 mm Offset; Test type: Superiority; p = .478, Kruskal-Wallis

6. Secondary Outcome: Oxford Shoulder Score (OSS) Questionnaire
Description: The Oxford Shoulder Score (OSS) is a patient reported questionnaire that includes 12 descriptors of pain and disability for shoulder ailments and related quality of daily activities. Each descriptor rating ranges from 0 to 4, with 4 representing the best (no pain, no difficulty with activity) and 0 is the worst (unbearable pain, extreme difficulty with activity). The score is calculated from the summation of all 12 descriptors, for a total range of 0 to 48, where a higher score reflects the best outcome (less pain and difficulty with activity) and a lower score reflects a worse outcome (more pain and difficulty with activity).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
Number analyzed (Participants) | 34 | 28 | 29 | 22
score on a scale | 6.8 (14.8) | 4.2 (8.9) | 11.0 (20.4) | 0.7 (0.1)
Statistical Analysis 1: Comparison: Small-Diameter Glenosphere +2 mm Offset vs Small-Diameter Glenosphere +6 mm Offset vs Large-Diameter Glenosphere +2 mm Offset vs Large-Diameter Glenosphere +6 mm Offset; Test type: Superiority; p = .527, ANOVA

7. Secondary Outcome: American Shoulder and Elbow Surgeons (ASES) Questionnaire
Description: A self-assessment that measures pain and ability to perform daily activities.The questionnaire is divided into 2 components, a single pain question and 10 questions on function of daily living.The total score is weighted 50% for pain and 50% for function. Pain is ranked from 0-10, where 0 is no pain and 10 is unbearable pain.The total pain score is calculated by subtracting the result of this question from 10 and multiplying by 5.The function score is calculated from the sum of 10 questions on daily living.The 10 questions are scored from 0-3, where 0=unable to perform daily activity and 3=no difficulty with daily activity.The individual function scores are summed for a maximum functional score of 30.This functional score is then multiplied by 5/3 to make the maximum functional score out of 50 possible points.The pain and function scores are then added together to obtain the final score out of 100.The final score ranges from 0 to 100, where higher scores correlate to better outcomes.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
Number analyzed (Participants) | 34 | 28 | 29 | 22
score on a scale | 50.7 (37.8) | 46.7 (39.5) | 56.8 (37.6) | 56.4 (35.6)
Statistical Analysis 1: Comparison: Small-Diameter Glenosphere +2 mm Offset vs Small-Diameter Glenosphere +6 mm Offset vs Large-Diameter Glenosphere +2 mm Offset vs Large-Diameter Glenosphere +6 mm Offset; Test type: Superiority; p = .823, ANOVA

8. Secondary Outcome: Quick DASH (Disabilities of the Arm Shoulder and Hand) Questionnaire
Description: The Quick DASH (disabilities of the arm, shoulder and hand) questionnaire is an 11 item self-reported participant questionnaire that measures physical function and symptoms in individuals experiencing musculoskeletal disorders of the upper limb. Each item is scored 1-5 where 1 reflects no pain or difficulty with activities and 5 reflects extreme pain or difficulty with activities. All individual scores are then summed and averaged to produce a score out of five. The score is then transformed to a score out of 100 by subtracting one and multiplying by 25. The final score ranges from 0 to 100, where a higher resulting score reflects more pain and greater disability while a lower score reflects less pain and disability.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
Number analyzed (Participants) | 34 | 28 | 29 | 22
score on a scale | 9.7 (0.6) | 9.1 (1.4) | 9.3 (1.4) | 8.3 (2.1)
Statistical Analysis 1: Comparison: Small-Diameter Glenosphere +2 mm Offset vs Small-Diameter Glenosphere +6 mm Offset vs Large-Diameter Glenosphere +2 mm Offset vs Large-Diameter Glenosphere +6 mm Offset; Test type: Superiority; p = .231, ANOVA

9. Secondary Outcome: Shoulder Pain
Description: Shoulder pain values reported by participants will be assessed using the 10cm Visual Analogue Scale (VAS). The VAS line will be 10 cm long with two endpoints representing 0 (no pain) and 10 (worst possible pain). Participants will identify their pain level by indicating a point on the line between each end. That point will be measured from the "No pain" end, and the number of centimeters will be reported as the pain score.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
Number analyzed (Participants) | 34 | 28 | 29 | 22
score on a scale | 0.3 (0.9) | 0.5 (0.9) | 0.3 (0.9) | 0.3 (0.8)
Statistical Analysis 1: Comparison: Small-Diameter Glenosphere +2 mm Offset vs Small-Diameter Glenosphere +6 mm Offset vs Large-Diameter Glenosphere +2 mm Offset vs Large-Diameter Glenosphere +6 mm Offset; Test type: Superiority; p = .595, Kruskal-Wallis

10. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with the outcome of the surgery measured by on a scale from 1-10, where 1 is not at all satisfied and 10 is very satisfied.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
Number analyzed (Participants) | 34 | 28 | 29 | 22
score on a scale | 9.6 (0.7) | 9.4 (1.0) | 9.2 (1.6) | 9.4 (0.8)
Statistical Analysis 1: Comparison: Small-Diameter Glenosphere +2 mm Offset vs Small-Diameter Glenosphere +6 mm Offset vs Large-Diameter Glenosphere +2 mm Offset vs Large-Diameter Glenosphere +6 mm Offset; Test type: Superiority; p = .789, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse events were collected on all participants from enrollment until approximately two years after surgery, for a total of approximately five years.
Arm/Group | Small-Diameter Glenosphere +2 mm Offset | Small-Diameter Glenosphere +6 mm Offset | Large-Diameter Glenosphere +2 mm Offset | Large-Diameter Glenosphere +6 mm Offset
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/28 | 0/29 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/34 | 5/28 | 0/29 | 0/22
Other Adverse Events (participants affected / at risk) | 0/34 | 3/28 | 0/29 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Small-Diameter Glenosphere +2 mm Offset (N=34) | Small-Diameter Glenosphere +6 mm Offset (N=28) | Large-Diameter Glenosphere +2 mm Offset (N=29) | Large-Diameter Glenosphere +6 mm Offset (N=22)
Reoperation (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Revision surgery (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Small-Diameter Glenosphere +2 mm Offset (N=34) | Small-Diameter Glenosphere +6 mm Offset (N=28) | Large-Diameter Glenosphere +2 mm Offset (N=29) | Large-Diameter Glenosphere +6 mm Offset (N=22)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Instability requiring modular component exchange (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Component failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT02768597/Prot_SAP_000.pdf